CLINICAL TRIAL: NCT05683951
Title: Phase III Clinical Trial to Evaluate the Efficacy and Safety of DWKH
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of DWKH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DWKH-302
Record Dates: First submitted 2022-05-30; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DWKH (Experimental)
  Interventions: Drug: DWKH
- DWKH-R (Active Comparator)
  Interventions: Drug: DWKH-R
- PLACEBO (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWKH — Administration of DWKH three times daily
  Arms: DWKH
Drug: DWKH-R — Administration of DWKH-R three times daily
  Arms: DWKH-R
Drug: Placebo — Administration of Placebo three times daily
  Arms: PLACEBO

SUMMARY:
Randomized, Double-blind, Parellel, Multicenter, Active-controlled

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged between 19 and 80.
* Patients whose BSS score is over 5.

Exclusion Criteria:

* Patients allergic to any ingredients of the study drugs.
* Moderate liver disease (ALT or AST > UNLx3).
* Moderate lung disease.
* Uncontrolled HTN.
* Uncontrolled DM.
* Uncontrolled thyroidism.
* Patients who is needed antibiotics during the study period.
* In the case of women, pregnant(Urine-HCG positive) or lactating women.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Bronchitis severity score (BSS) | 0,4,7 days
  Difference of the BSS score (0 to 4, higher score means more severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea